CLINICAL TRIAL: NCT05205213
Title: Stepwise for the Treatment of Lateral Incisional Hernias
Status: Completed | Type: Observational
Sponsor: Henares University Hospital (Other)
Responsible Party: Principal Investigator, Miguel A ngel Garci-a Urena, Head of General Surgery Service, Henares University Hospital
Other Study IDs: 39/2019.
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Incisional Hernia; Abdominal Wall Defect; Abdominal Wall Hernia; Hernia
MeSH Terms: conditions — Incisional Hernia; Hernia, Abdominal; Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lateral retromuscular preperitoneal group: All patients undergoing open lateral retromuscular preperitoneal repair through the previous lateral incision for L3-L4 IHs between February 2012 and January 2020
  Interventions: Other: Surgical Technique (lateral retromuscular preperitoneal)
- Reverse TAR group: All patients undergoing open reverse TAR repair through the previous lateral incision for L3-L4 IHs between February 2012 and January 2020

INTERVENTIONS:
Other: Surgical Technique (lateral retromuscular preperitoneal) — Open abdominal wall repair through the previous lateral incision for L3-L4 Incisional hernias
  Other Names: Surgical Technique (reverse TAR)
  Groups: lateral retromuscular preperitoneal group

SUMMARY:
The best approach for lateral incisional hernia is not known. Posterior component separation (reverse TAR) offers the possibility of using the retromuscular space for medial extension of the challenging preperitoneal plane.

The main objective of the study was to describe the surgical techniques used and their outcomes in the open lateral approach for the treatment of L3-L4 European Hernia Society (EHS) classification Incisional hernias, comparing the results between reverse TAR and pure lateral retromuscular preperitoneal, and analyzing the short- and long- term complications, including patient-reported outcomes measures (PROMs).

The study report followed the recommendations for reporting outcomes in abdominal wall hernias, and the new international classification of abdominal wall planes (ICAP).

A multicenter retrospective observational study was conducted using a prospectively maintained database from three university hospitals in Spain specialized in complex abdominal wall reconstruction. All patients undergoing open abdominal wall repair through the previous lateral incision for L3-L4 IHs between February 2012 and January 2020 were identified. All patients were operated on by the senior surgeons responsible for the complex abdominal wall units of each participating center. Prior to conducting the study, the approval of the local ethics committee was obtained (ID:39/2019). Written informed consent was also obtained.

The diagnosis of IH was based on clinical examination and imaging from a computed tomography (CT). The investigator only included patients with L3-L4 IHs. Patients with primary lateral hernias, such as Spiegel, Grynfelt and Petit hernias were excluded. We also excluded all patients in which the lateral IH was a parastomal hernia.

Demographic data, patient comorbidities, different classifications of hernia complexity, Carolinas Equation for Determining Associated Risks (CeDAR) and intraoperative and postoperative data were collected All patients followed a similar preoperative optimization program, which included endocrinologic and nutritional evaluations, respiratory physiotherapy, and abstinence from smoking at least 1 month before surgery. Weight loss was extremely recommended but without any mandatory prerequisite.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a lateral incisional hernia L3 European Hernia Society classification
* Patients with a lateral incisional hernia L4 European Hernia Society classification
* Patients older than 18 years old

Exclusion Criteria:

* Midline incisional hernia.
* Patients with a parastomal hernia
* Patients with a primary midline ventral hernia
* Patients with a primary lateral hernia.
* Age under 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing open abdominal wall repair through the previous lateral incision for L3-L4 IHs between February 2012 and January 2020 in the three University Hospitals in Spain involving in the multicentric study
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2012-02-06 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Recurrence | At least 12 month
  Recurrence was defined as a bulge of the contents of the abdominal cavity or preperitoneal fat through an abdominal wall defect at the site of a previous abdominal wall hernia repair.

SECONDARY OUTCOMES:
Surgical Site Occurrence | 30 days
  Surgical Site Occurrence: the definition standardized by the Ventral Hernia Working Group (VHWG) was used, which includes any SSI, and wound cellulitis, unhealed incisional wound, fascial disruption, skin or soft tissue ischemia, skin or soft tissue necrosis, serous or purulent drainage wound, suture abscess, seroma, hematoma, infected or exposed mesh, or development of an enterocutaneous fistula
Surgical Site Occurrence Requiring Procedural Intervention (SSOPI) | 30 days
  Surgical Site Occurrence Requiring Procedural Intervention (SSOPI): any SSO requiring wound opening, wound debridement, suture removal, percutaneous drainage, or partial or complete removal of the mesh
Surgical Site Infection (SSI) | 30 days
  Surgical Site Infection (SSI) was defined using the standardized CDC definition: "infection that occurs in the part of the body where surgery has been performed and includes superficial, deep, and organ / space types"
Bulging | At least 12 month
  Bulging was defined as an area of weakness or asymmetry on inspection or exploration of the patient's abdominal wall, with no confirmed defects on CT.
European Registry for Abdominal Wall Hernias Quality of Life scale ("EuraHS-QoL") | 24 months
  Quality of life study was developed using the "European Registry for Abdominal Wall Hernias Quality of Life" scale ("EuraHS-QoL"), a specific tool developed by the EHS, which compares the evolution of the patients between the preoperative and postoperative periods regarding pain, restriction and aesthetic appearance domains. The minimum value is 0 and maximum value is 10. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel Angel Garcia Ureña, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We want to protect all the personal data of the patients participating in the study

REFERENCES:
- [Background] Parker SG, Halligan S, Liang MK, Muysoms FE, Adrales GL, Boutall A, de Beaux AC, Dietz UA, Divino CM, Hawn MT, Heniford TB, Hong JP, Ibrahim N, Itani KMF, Jorgensen LN, Montgomery A, Morales-Conde S, Renard Y, Sanders DL, Smart NJ, Torkington JJ, Windsor ACJ. International classification of abdominal wall planes (ICAP) to describe mesh insertion for ventral hernia repair. Br J Surg. 2020 Feb;107(3):209-217. doi: 10.1002/bjs.11400. Epub 2019 Dec 25. PMID 31875954
- [Background] Haskins IN, Horne CM, Krpata DM, Prabhu AS, Tastaldi L, Perez AJ, Rosenblatt S, Poulose BK, Rosen MJ. A call for standardization of wound events reporting following ventral hernia repair. Hernia. 2018 Oct;22(5):729-736. doi: 10.1007/s10029-018-1748-6. Epub 2018 Feb 10. PMID 29429064
- [Background] Garner JS. CDC guideline for prevention of surgical wound infections, 1985. Supersedes guideline for prevention of surgical wound infections published in 1982. (Originally published in November 1985). Revised. Infect Control. 1986 Mar;7(3):193-200. doi: 10.1017/s0195941700064080. No abstract available. PMID 3633903
- [Background] Muysoms F, Campanelli G, Champault GG, DeBeaux AC, Dietz UA, Jeekel J, Klinge U, Kockerling F, Mandala V, Montgomery A, Morales Conde S, Puppe F, Simmermacher RK, Smietanski M, Miserez M. EuraHS: the development of an international online platform for registration and outcome measurement of ventral abdominal wall hernia repair. Hernia. 2012 Jun;16(3):239-50. doi: 10.1007/s10029-012-0912-7. Epub 2012 Apr 18. PMID 22527930
- [Result] Muysoms FE, Miserez M, Berrevoet F, Campanelli G, Champault GG, Chelala E, Dietz UA, Eker HH, El Nakadi I, Hauters P, Hidalgo Pascual M, Hoeferlin A, Klinge U, Montgomery A, Simmermacher RK, Simons MP, Smietanski M, Sommeling C, Tollens T, Vierendeels T, Kingsnorth A. Classification of primary and incisional abdominal wall hernias. Hernia. 2009 Aug;13(4):407-14. doi: 10.1007/s10029-009-0518-x. Epub 2009 Jun 3. PMID 19495920
- [Result] Muysoms FE, Deerenberg EB, Peeters E, Agresta F, Berrevoet F, Campanelli G, Ceelen W, Champault GG, Corcione F, Cuccurullo D, DeBeaux AC, Dietz UA, Fitzgibbons RJ Jr, Gillion JF, Hilgers RD, Jeekel J, Kyle-Leinhase I, Kockerling F, Mandala V, Montgomery A, Morales-Conde S, Simmermacher RK, Schumpelick V, Smietanski M, Walgenbach M, Miserez M. Recommendations for reporting outcome results in abdominal wall repair: results of a Consensus meeting in Palermo, Italy, 28-30 June 2012. Hernia. 2013 Aug;17(4):423-33. doi: 10.1007/s10029-013-1108-5. Epub 2013 May 15. PMID 23673408